CLINICAL TRIAL: NCT01418768
Title: Effects of an Inpatient Rehabilitation for Patients With Chronic Obstructive Pulmonary Disease (COPD) III/IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician pneumology, Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT2011
Record Dates: First submitted 2011-08-09; First posted 2011-08-17 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; CAT; Rehabilitation; chronic obstructive pulmonary disease GOLD III/IV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rehabilitation (Experimental)
  Interventions: Other: inpatient rehabiliation

INTERVENTIONS:
Other: inpatient rehabiliation — inpatient, multimodal, individual workout including endurance training, strength training, coordination training etc. for three weeks.

SUMMARY:
The purpose of this study is to determine if there is a change in the CAT-score after an inpatient rehabilitation of three weeks and if it correlates with other common parameters.

ELIGIBILITY:
Inclusion Criteria:

* inpatient rehabilitation in Schön Klinik Berchtesgadener Land
* stable COPD(GOLD severity III and IV with and without respiratory insufficiency)

Exclusion Criteria:

* severe exacerbation in the last four weeks
* acute coronary syndrome
* unability to cooperate

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in CAT-score | day 1 to day 21

SECONDARY OUTCOMES:
Change in 6 minutes walking distance | day 1 to day 21
Change in Short-Form 36 | day 1 to day 21
Change in Hospital Anxiety and Depression Scale | day 1 to day 21
Change in diffusing capacity | day 1 to day 21
Change in forced expiratory volume in 1 second (FEV1) | day 1 to day 21
Change in Body Mass index | day 1 to day 21
Change in basal energy rate | day 1 to day 21
Change in BODE-Index | day 1 to day 21
Change in St. George's Respiratory Questionaire | Day 1 to day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany